CLINICAL TRIAL: NCT02038062
Title: Influence of Sevoflurane Preconditioning on Tissue Oxygenation of the Tibial Anterior Muscle Measured by Near-infrared Spectroscopy After Clamping of the Femoral Artery for Vascular Surgery
Brief Title: Tissue Oxygenation of the Tibial Anterior Muscle After Clamping of the Femoral Artery
Acronym: NIRSFEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Axel Fudickar, Dr., University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Fudickar7
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Tissue Oxygen Saturation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevoflurane (Experimental): Sevoflurane Preconditioning
  Interventions: Procedure: Sevoflurane preconditioning
- No Sevoflurane (No Intervention): No Sevoflurane Preconditioning

INTERVENTIONS:
Procedure: Sevoflurane preconditioning — Preconditioning by transient application of sevoflurane
  Arms: Sevoflurane

SUMMARY:
Ischemic preconditioning is defined as protection from cell damage induced by prolonged ischemia by preceding cycles of short ischemia. Hence, ischemic preconditioning could reduce ischemic lesion during clamping a femoral artery for vascular surgery. In this prospective, randomized pilot study is investigated if clamping of the femoral artery leads to ischemia of the calf measurable by near-infrared spectroscopy. In addition to this, the effect of sevoflurane preconditioning on ischemia of the calf is measured.

DETAILED DESCRIPTION:
Ischemic preconditioning is performed by clamping of the femoral artery for five minutes in 40 patients. In 20 patients sevoflurane preconditioning is performed five minutes before ischemic preconditioning by inducing sevoflurane anesthesia for five minutes. Muscle tissue oxygenation is measured bilaterally in the anterior tibial muscle by near-infrared spectroscopy (INVOS, SOMANETICS, Troy, Michigan/ USA) during preconditioning and following ischemia.Clinically relevant ischemia was defined as a decrease of tissue oxygen saturation to 95 % of baseline.

ELIGIBILITY:
Inclusion Criteria:vascular surgery with clamping of a femoral artery. -

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Decrease of tissue oxygen saturation below 95 % of baseline | 4 hours
  Decrease of tissue oxygen saturation below 95 % of baseline

CONTACTS AND LOCATIONS:
Overall Officials: Axel Fudickar, Dr., Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein, Germany

REFERENCES:
- [Derived] Fudickar A, Kunath S, Voss D, Siggelkow M, Cavus E, Steinfath M, Bein B. Effect of ischemic and pharmacological preconditioning of lower limb muscle tissue on tissue oxygenation measured by near-infrared spectroscopy--a pilot study. BMC Anesthesiol. 2014 Jul 15;14:54. doi: 10.1186/1471-2253-14-54. eCollection 2014. PMID 25132803